CLINICAL TRIAL: NCT05701644
Title: A Dose-block Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose, First-in-human, Phase 1 Clinical Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics After Subcutaneous Administration of C1K in Healthy Subjects
Brief Title: Study To Evaluate the Safety, Tolerability, and Pharmacokinetics After Subcutaneous Administration of C1K in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ensol Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C1K-101
Record Dates: First submitted 2022-12-22; First posted 2023-01-27 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2023-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- C1K 150mg (Experimental): Subcutaneous Administration C1K 150mg single or multi dose
  Interventions: Drug: C1K 150mg
- C1K 300mg or placebo (Experimental): Subcutaneous Administration C1K 300mg or placebo single or multi dose
  Interventions: Drug: C1K 300mg; Drug: Placebo with the same volume of C1K 300mg
- C1K 600mg or placebo (Experimental): Subcutaneous Administration C1K 600mg or placebo single or multi dose
  Interventions: Drug: C1K 600mg; Drug: Placebo with the same volume of C1K 600mg
- C1K 900mg or placebo (Experimental): Subcutaneous Administration C1K 900mg or placebo single or multi dose
  Interventions: Drug: C1K 900mg; Drug: Placebo with the same volume of C1K 900mg
- C1K 1200mg or placebo (Experimental): Subcutaneous Administration C1K 1200mg or placebo single or multi dose
  Interventions: Drug: C1K 1200mg; Drug: Placebo with the same volume of C1K 1200mg

INTERVENTIONS:
Drug: C1K 150mg — Subcutaneously administrate C1K 150mg at Day 1, Day 8, Day 15
  Arms: C1K 150mg
Drug: C1K 300mg — Subcutaneously administrate C1K 300mg at Day 1, Day 8, Day 15
  Arms: C1K 300mg or placebo
Drug: Placebo with the same volume of C1K 300mg — Subcutaneously administrate placebo with the same volume of C1K 300mg at Day 1, Day 8, Day 15
  Arms: C1K 300mg or placebo
Drug: C1K 600mg — Subcutaneously administrate C1K 600mg at Day 1, Day 8, Day 15
  Arms: C1K 600mg or placebo
Drug: Placebo with the same volume of C1K 600mg — Subcutaneously administrate placebo with the same volume of C1K 600mg at Day 1, Day 8, Day 15
  Arms: C1K 600mg or placebo
Drug: C1K 900mg — Subcutaneously administrate C1K 900mg at Day 1, Day 8, Day 15
  Arms: C1K 900mg or placebo
Drug: Placebo with the same volume of C1K 900mg — Subcutaneously administrate placebo with the same volume of C1K 900mg at Day 1, Day 8, Day 15
  Arms: C1K 900mg or placebo
Drug: C1K 1200mg — Subcutaneously administrate C1K 1200mg at Day 1, Day 8, Day 15
  Arms: C1K 1200mg or placebo
Drug: Placebo with the same volume of C1K 1200mg — Subcutaneously administrate placebo with the same volume of C1K 1200mg at Day 1, Day 8, Day 15
  Arms: C1K 1200mg or placebo

SUMMARY:
A dose-block randomized, double-blind, placebo-controlled, single and multiple ascending dose, first-in-human, phase 1 first in human clinical trial to evaluate the safety, tolerability, and pharmacokinetics after subcutaneous administration of C1K in healthy Korean subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects aged 19 - 45 years at the time of screening visit procedure.
2. The subject weighs in the range of 50.0 - 90.0 kg and has a body mass index (BMI) in the range 18-27 kg/m2.
3. Sufficient ability to understand the study after being informed about the study and provide written informed consent.
4. Based on physical examination, vital sign, 12-lead ECG and laboratory test etc. and in the opinion of the investigator, the subject is suitable for the study.

Exclusion Criteria:

1. A subject with clinically significant hepatobiliary, renal, neurologic, respiratory, endocrine, blood•oncology, cardiovascular, urinary, or, psychical diseases or a history
2. A subject who has difficulty with sub-cutaneous injection(ex: tattoo, allergy on skin etc.)
3. A subject who has hypersensitivity to the drugs of the drugs containing the same class, or other drugs, or a history of clinically significant hypersensitivity
4. A subject who has ventricular tachycardia, ventricular tachycardia, ventricular flutter or confirmed other ventricular flutter and QTc interval: > 450 ms or the other clinically significant medical findings
5. A subject with the following results in the screening test:

   * Blood AST (GOT), ALT (GPT): > Normal range upper × 1.5
   * Blood CPK > Normal range upper × 1.5
   * eGFR (CKD-EPI equation) < 60 mL/min/1.73 m2
6. Positive serological test (syphilis test, hepatitis B test, hepatitis C test, human immunodeficiency virus (HIV) test)
7. A subject with the following results in the screening test:

   * systolic blood pressure < 80 mmHg or > 140 mmHg
   * diastolic blood pressure < 50 mmHg or > 90 mmHg
8. A subject with a history of drug abuse or positive urine screening test for drug abuse
9. A subject who administered any prescription drugs or herbal medicine within 2 weeks prior to the expected date of the first dose, or any over-the-counter drug (OTC drug) or vitamin within 1 week prior to the expected date of the first dose (However, can participate in the study if otherwise decided eligible by the investigator).
10. A subject who participated in other clinical trial and administered investigational drug within 6 months prior to the expected date of the first dose
11. A subject who donated whole blood within 2 months or the component blood within 1 month prior to the expected date of the first dose, or received blood transfusion within 1 month prior to the expected date of the first dose
12. Smokers who smoke more than 10 cigarettes/day in the last 3 months as of screening day.
13. A subject with persistent alcohol intake (> 21 units/week, 1 unit = 10 g of pure alcohol), or inability to abstain from drinking from 3 days before the expected date of the first dose until the last discharge
14. A male subject who has plan to have a baby or to donate sperm. A female subject who is pregnant or lactating or has plan to lactate within 3 months after administration of IP
15. A subject who is intending to become pregnant during this study or with inability to use a medically acceptable contraception method(ex. sterilization operation, intrauterine device etc. for Subject or subject's partner

    ※ medically acceptable contraception method
    * Use of intrauterine device which is proven pregnancy failure rates in spouses (or partners).
    * Use combined blocking contraceptives (for male or female) and antiseptic drugs
    * Subject or partner's operation(vasectomized, bilateral tubal occlusion, hysterectomy)
16. Subject who is considered inadequate to participation in the study due to other reason under investigator's discretion

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability Assessment | Day -1 to Day 23
  Percentage of occurrences observed Adverse Event in each group.
Safety and Tolerability Assessment by Value Changes in Vital Signs | Day -1 to Day 23
  Vital Signs including blood pressure and heart rate changes from baseline.
Safety and Tolerability Assessment by Value Changes in Physical Examination | Day -1 to Day 23
  physical examination changes from baseline.
Safety and Tolerability Assessment by Value Changes in Laboratory Test | Day -1 to Day 23
  laboratory test changes from baseline assessed through hematology, blood biochemistry, urinalysis and blood coagulation.
Safety and Tolerability Assessment by Value Changes in 12-Lead Electrocardiogram | Day -1 to Day 23
  12-Lead Electrocardiogram(ECG) changes from baseline.
Safety and Tolerability Assessment by Response Change of Injection site. | Day 1 to Day 23
  Percentage of occurrences observed response change of injection site.
Pharmacokinetic Assessment by Maximum concentration of C1K in plasma | Day 1/ Day 15 pre-dose(0 hour), 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hour at Day 1 and Day 15
  Maximum concentration of C1K in plasma (Cmax)
Pharmacokinetic Assessment by Area Under the Plasma Concentration-Time Curve of C1K from Time Zero to the Last Measurable Point | Day 1/ Day 15 pre-dose(0 hour), 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hour at Day 1 and Day 15
  Area under the plasma C1K concentration-time curve from 0 to last(AUClast)
Pharmacokinetic Assessment by Area under the plasma C1K concentration-time curve from 0 to infinity | Day 1/ Day 15 pre-dose(0 hour), 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hour at Day 1 and Day 15
  Area under the plasma C1K concentration-time curve from 0 to last(AUCinf)
Pharmacokinetic Assessment by The time of peak concentration of C1K | Day 1/ Day 15 pre-dose(0 hour), 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hour at Day 1 and Day 15
  The time of peak concentration(Tmax)
Pharmacokinetic Assessment by Elimination half-life of C1K | Day 1/ Day 15 pre-dose(0 hour), 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hour at Day 1 and Day 15
  Elimination half-life(t1/2)
Pharmacokinetic Assessment by Apparent Clearance of C1K | Day 1/ Day 15 pre-dose(0 hour), 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hour at Day 1 and Day 15
  Apparent Clearance(CL/F)
Pharmacokinetic Assessment by Apparent Volume of Distribution After extravascular administration of C1K | Day 1/ Day 15 pre-dose(0 hour), 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hour at Day 1 and Day 15
  Apparent Volume of Distribution After extravascular administration(Vz/F)
Pharmacokinetic Assessment by Accumulation Ratio of C1K | Day 1/ Day 15 pre-dose(0 hour), 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hour at Day 1 and Day 15
  Accumulation Ratio(Rac)
Pharmacokinetic Assessment by Minimum concentration of C1K in plasma | Day 1/ Day 15 pre-dose(0 hour), 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hour at Day 1 and Day 15
  Minimum concentration of C1K in plasma(Cmin,ss)
Pharmacokinetic Assessment by Average concentration of C1K in plasma | Day 1/ Day 15 pre-dose(0 hour), 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hour at Day 1 and Day 15
  Average concentration of C1K in plasma(Cav)
Pharmacokinetic Assessment by Peak to trough fluctuation ratio | Day 1/ Day 15 pre-dose(0 hour), 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hour at Day 1 and Day 15
  Peak to trough fluctuation ratio(PTF)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No